CLINICAL TRIAL: NCT05129917
Title: The Anti-fatigue Effect of Gojinsen® Drink
Brief Title: Effects of Supplementation With Ginseng and BCAA Improved Central Fatigue and Enhanced Attention During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSMH No.13-023-A2
Record Dates: First submitted 2021-11-11; First posted 2021-11-22 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Exercise Addiction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): consume 1 sachet per day for 14 day
  Interventions: Dietary Supplement: Placebo
- Gojinsen® drinks (Experimental): consume 1 sachet per day for 14 day
  Interventions: Dietary Supplement: Gojinsen® drinks

INTERVENTIONS:
Dietary Supplement: Placebo — consume 1 sachet per day for 14 day
  Arms: Placebo
Dietary Supplement: Gojinsen® drinks — consume 1 sachet per day for 14 day
  Arms: Gojinsen® drinks

SUMMARY:
The main purpose of the present study is to determine the effects of acute and short-term (14 days) ginseng combined with branch chained amino acids supplementation on endurance exercise performance and the ability of anti-fatigue. In addition, this study also measured the performance of continuous attention during recovery period to examine the effect of supplementation on central fatigue.

DETAILED DESCRIPTION:
Muscle fatigue was a common problem after exercise. When fatigue occured, body functions were affected and changed. Changbai Mountain ginseng had higher anti-fatigue substances than general commercial ginseng. And recent studies had showed that the supplementation of branched chain amino acids (BCAA), including leucine, isoleucine and valine, can increase attention and reduce fatigue. However, its effect on Changbai Mountain ginseng combined with BCAA was still unclear. Subjects were allocated to Gojinsen® drinks and placebo group (1:1 ratio) for 14 days, and then examined by maximal oxygen consumption, time to exhaustion, rating of perceived exertion (RPE), oxygen saturation (SPO2) , blood lactate concentration, and continuous attention performance test (CPT II). The Gojinsen® group significant increased maximal oxygen consumption, time to exhaustion, and attention compared to placebo group. Moreover, the Gojinsen® group significant decreased lactate concentration and fatigue compared to placebo group. By this study, Gojinsen® drinks did not showed absolute anti-fatigue effect but provided the objective evidence of fatigue-related measurement and the therapeutic potential for people suffering from exercise fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. healthy male and female adults aged 20-25 years old .
2. without heart, liver, kidney, endocrine or other major organic diseases).
3. had at least 3 months experience in performing exercise

Exclusion Criteria:

1. BMI of the study subjects must be less than 25.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Endurance exercise performance testing | Execution on the 14th day
  the subjects arrived to the laboratory and wore the oxygen uptake mask of energy metabolism analyzer (Sensor Medics, Vmax29, USA) to measure the subjects' oxygen uptake
rating of perceived exertion | Execution on the 14th day
  The Rated Perceived Exertion was measured during the treadmill exercise by Bruce Protocol, a gradual increase in the speed and the slope of the treadmill every 3 minutes.
blood lactate | Execution on the 14th day
  fingertip capillary blood was placed in automated blood lactate analyzer
Continuous attention performance test | Execution on the 14th day
  10 minutes after maximal exercise test, the subjects performed attention tests that used Canon continuous attention software

CONTACTS AND LOCATIONS:
Overall Officials: Bo han Wu, Ph.D, Principal Investigator — Pingtung University of Science and Technology